CLINICAL TRIAL: NCT01825798
Title: Treatment of Overweight Induced by Antipsychotic Medication in Young People With Autism Spectrum Disorders (ASD)
Acronym: MET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Vanderbilt University (Other); University of Pittsburgh Medical Center (Other); Nationwide Children's Hospital (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET-10-2012
Record Dates: First submitted 2013-02-07; First posted 2013-04-08 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2018-01

CONDITIONS: Overweight; Autism Spectrum Disorder
Keywords: Metformin; Overweight; Atypical Antipsychotic; Medication; Randomized Clinical Trial; Children
MeSH Terms: conditions — Overweight; Autism Spectrum Disorder | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Hydrochloride Oral Solution (Placebo Comparator)
  Interventions: Drug: Placebo
- Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin will be dispensed in a liquid suspension of 100 mg/mL. For children 6-9 years of age, metformin will be started at 250 mg at their evening meal for 1 week, followed by the addition of a 250 mg dose at breakfast for 1 week. At the Week 2 visit, if metformin is well-tolerated, the dose will be increased to 500 mg twice daily. For children from 10-17 years of age, metformin will be started at 250 mg at their evening meal for 1 week, followed by the addition of a 250 mg dose at breakfast for 1 week. At the Week 2 visit, if metformin is well-tolerated, the dose will be increased to 500 mg twice daily. At the Week 4 visit, if metformin is well-tolerated, the dose will be increased to 850 mg twice daily.
  Other Names: Riomet
  Arms: Metformin
Drug: Placebo — The placebo hydrochloride oral solution will be prepared to match the appearance, smell and taste of the metformin as closely as possible. For children from 6-9 years of age, placebo will be started at 250 mg at their evening meal for 1 week, followed by the addition of a 250 mg dose at breakfast for 1 week. At the Week 2 visit, if placebo is well-tolerated, the dose will be increased to 500 mg twice daily. For children from 10-17 years of age, placebo will be started at 250 mg at their evening meal for 1 week, followed by the addition of a 250 mg dose at breakfast for 1 week. At the Week 2 visit, if placebo is well-tolerated, the dose will be increased to 500 mg twice daily. At the Week 4 visit, if placebo is well-tolerated, the dose will be increased to 850 mg twice daily.
  Arms: Placebo Hydrochloride Oral Solution

SUMMARY:
The purpose of this study is to determine whether metformin is safe and effective in the treatment of weight or weight gain in young people with Autism Spectrum Disorders (ASD) who are currently taking atypical antipsychotic medication.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, multi-site randomized trial to evaluate oral fixed dose metformin (Riomet®) in decreasing weight or weight gain in children ages 6-17 years, 4 months with ASD who are currently taking atypical antipsychotic medication. A 16-week, double-blind, placebo-controlled randomized trial of metformin with dose guided by age will be conducted. A secondary study aim will be to assess the long-term safety and efficacy of metformin by conducting a 16-week open label continuation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Autism Spectrum Disorder (autistic disorder, pervasive developmental disorder not otherwise specified), Asperger's disorder) based upon an Autism Diagnostic Observation Scale (ADOS) and Diagnostic and Statistical Manual (DSM-IV) interview.
2. Minimum of 1 month on a stable atypical antipsychotic dose with no plans to change the dose for the next 4 months.
3. A documented greater than/equal to 7% increase in BMI since starting atypical antipsychotic therapy(going back as far as prior 12 months); or, if BMI is greater or equal to 85th percentile corrected for age and sex, then a greater than 5% body weight increase per year (prorated at greater than 5% body weight increase if medicated for longer than a year).
4. Age 6 years to 17 years, 4 months.
5. Subjects and their parents (guardians) must be judged reliable for medication compliance and must agree to keep appointments for study visits and tests as outlined in the protocol.
6. Prior to the conduct of any study-specific procedures, the subject must provide assent to participate in the study (if developmentally appropriate), and their parents (guardians) must provide written informed consent.

Exclusion Criteria:

1. History of intolerable adverse effects with metformin.
2. Prior history of an exposure to metformin of sufficient dose or duration to determine response status.
3. History of liver disease, renal impairment, congestive heart failure, pernicious anemia, any other condition increasing the risk for lactic acidosis, or any serious medical illness requiring treatment.
4. Use of cationic drugs excreted by the kidneys.
5. Planned surgery or procedure requiring contrast.
6. Pregnant at screening contact.
7. On other psychotropic concomitant medications for less than 2 months.
8. Treatment or planned treatment with concomitant medications with unacceptable interactions with metformin, including topiramate, levetiracetam, beta blockers, angiotensin-converting-enzyme (ACE) inhibitors, diuretics, or histamine H2 receptor antagonists.
9. Unable to tolerate blood work.
10. Current use of medication for target symptoms of appetite or weight loss.
11. Planned change of medication, medication dose, or behavioral treatment targeting weight loss during the study period.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, M.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Jeremey Veenstra-VanderWeele, M.D., Principal Investigator — Columbia University; Benjamin Handen, Ph.D., Principal Investigator — University of Pittsburgh Medical Center; Michael Aman, Ph.D., Principal Investigator — Ohio State University/Nationwide Children's Hospital; Eric Butter, Ph.D., Principal Investigator — Nationwide Children's Hospital; Kevin Sanders, M.D., Principal Investigator — Vanderbilt University
Locations (4):
- United States (3):
  - Ohio State University/Nationwide Children's Hospital, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Handen BL, Anagnostou E, Aman MG, Sanders KB, Chan J, Hollway JA, Brian J, Arnold LE, Capano L, Williams C, Hellings JA, Butter E, Mankad D, Tumuluru R, Kettel J, Newsom CR, Peleg N, Odrobina D, McAuliffe-Bellin S, Marler S, Wong T, Wagner A, Hadjiyannakis S, Macklin EA, Veenstra-VanderWeele J. A Randomized, Placebo-Controlled Trial of Metformin for the Treatment of Overweight Induced by Antipsychotic Medication in Young People With Autism Spectrum Disorder: Open-Label Extension. J Am Acad Child Adolesc Psychiatry. 2017 Oct;56(10):849-856.e6. doi: 10.1016/j.jaac.2017.07.790. Epub 2017 Aug 19. PMID 28942807
- [Derived] Anagnostou E, Aman MG, Handen BL, Sanders KB, Shui A, Hollway JA, Brian J, Arnold LE, Capano L, Hellings JA, Butter E, Mankad D, Tumuluru R, Kettel J, Newsom CR, Hadjiyannakis S, Peleg N, Odrobina D, McAuliffe-Bellin S, Zakroysky P, Marler S, Wagner A, Wong T, Macklin EA, Veenstra-VanderWeele J. Metformin for Treatment of Overweight Induced by Atypical Antipsychotic Medication in Young People With Autism Spectrum Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Sep 1;73(9):928-37. doi: 10.1001/jamapsychiatry.2016.1232. PMID 27556593

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Started | 32 | 28
Completed | 30 | 23
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 5
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 28 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.7 (2.64) | 12.9 (2.85) | 12.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 24 | 21 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 29 | 28 | 57
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 28 | 22 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 8 | 16
  United States | 24 | 20 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index Z-score
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: 16-wk change in BMI z-score
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
16-wk change in BMI z-score | 0.02 [-0.03 to 0.06] | -0.08 [-0.13 to -0.04]

2. Secondary Outcome: Changes in Additional Body Composition Parameters (Absolute Change in Weight)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: 16-wk change in weight (kg)
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
16-wk change in weight (kg) | 2.80 [1.90 to 3.70] | 0.07 [-0.88 to 1.02]

3. Secondary Outcome: Changes in Additional Body Composition Parameters (Relative Change in Weight)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: 16-wk change in weight (z-score)
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
16-wk change in weight (z-score) | 0.04 [-0.01 to 0.08] | -0.10 [-0.15 to -0.05]

4. Secondary Outcome: Changes in Additional Body Composition Parameters (Absolute BMI)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: 16-wk change in BMI (kg/m2)
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
16-wk change in BMI (kg/m2) | 0.52 [0.18 to 0.87] | -0.43 [-0.80 to -0.06]

5. Secondary Outcome: Changes in Additional Body Composition Parameters (Abdominal Circumference)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: centimetres
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
centimetres | 1.45 [0.39 to 2.51] | -0.21 [-1.32 to 0.91]

6. Secondary Outcome: Changes in Additional Body Composition Parameters (Hip Circumference)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: centimetres
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
centimetres | 1.06 [-0.06 to 2.17] | -0.63 [-1.81 to 0.54]

7. Secondary Outcome: Changes in Fasting Metabolic Parameters (Total Cholesterol)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: 16-week change total cholesterol (mg/dL)
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
16-week change total cholesterol (mg/dL) | -3.29 [-10.33 to 3.75] | -1.05 [-8.76 to 6.67]

8. Secondary Outcome: Changes in Fasting Metabolic Parameters (LDL)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: 16-week change in LDL (mg/dL)
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
16-week change in LDL (mg/dL) | -0.41 [-6.11 to 5.29] | -4.41 [-10.47 to 1.64]

9. Secondary Outcome: Changes in Fasting Metabolic Parameters (HDL)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: 16-week change in HDL (mg/dL)
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
16-week change in HDL (mg/dL) | -0.98 [-5.26 to 3.29] | 3.27 [-1.41 to 7.94]

10. Secondary Outcome: Changes in Fasting Metabolic Parameters (Triglycerides)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: 16-week change in triglycerides (mg/dL)
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
16-week change in triglycerides (mg/dL) | 6.18 [-19.62 to 31.98] | 5.74 [-22.34 to 33.81]

11. Secondary Outcome: Changes in Fasting Metabolic Parameters (Glucose)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: 16-week change in gluclose (mg/dL)
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
16-week change in gluclose (mg/dL) | -2.41 [-5.76 to 0.94] | -3.06 [-6.68 to 0.56]

12. Secondary Outcome: Changes in Fasting Metabolic Parameters (Insulin)
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: 16-week change insulin fasting (µIU/mL)
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Number analyzed (Participants) | 32 | 28
16-week change insulin fasting (µIU/mL) | 2.95 [-8.44 to 14.35] | 1.97 [-10.44 to 14.38]

ADVERSE EVENTS:
Arm/Group | Placebo Hydrochloride Oral Solution | Metformin
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/28
Other Adverse Events (participants affected / at risk) | 32/32 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Hydrochloride Oral Solution (N=32) | Metformin (N=28)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) — history of hospital admission for aggression
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Hydrochloride Oral Solution (N=32) | Metformin (N=28)
Overall (Ear and labyrinth disorders) | 3 (4) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 3 (4) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal Pain, upper (Gastrointestinal disorders) | 4 (4) | 3 (3)
Abnormal Feces (Gastrointestinal disorders) | 0 (0) | 3 (3)
Chapped lips (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 13 (19) | 17 (26)
Flatulence (Gastrointestinal disorders) | 3 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (8) | 8 (9)
Overall (Gastrointestinal disorders) | 19 (55) | 24 (64)
Fatigue (General disorders) | 6 (6) | 6 (8)
Irritability (General disorders) | 7 (7) | 7 (9)
Product taste abnormal (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 1 (2) | 3 (4)
Overall (General disorders) | 14 (18) | 13 (27)
Ear Infection (Infections and infestations) | 1 (1) | 2 (4)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (4)
Otitis media (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 6 (6)
Overall (Infections and infestations) | 19 (25) | 14 (24)
Overall (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Blood insulin level increased (Investigations) | 2 (2) | 2 (2)
Blood triglyceride level increased (Investigations) | 2 (2) | 1 (1)
Overall (Investigations) | 5 (7) | 4 (4)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 8 (8)
Increased Appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Overall (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Overall (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (5)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 6 (9) | 5 (8)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2)
Overall (Nervous system disorders) | 10 (16) | 12 (20)
Affect Lability (Psychiatric disorders) | 4 (4) | 0 (0)
Aggression (Psychiatric disorders) | 2 (3) | 5 (6)
Anger (Psychiatric disorders) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Depressed Mood (Psychiatric disorders) | 2 (2) | 0 (0)
Initial Insomnia (Psychiatric disorders) | 2 (3) | 3 (3)
Middle Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Overall (Psychiatric disorders) | 13 (27) | 14 (27)
Overall (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Overall (Respiratory, thoracic and mediastinal disorders) | 12 (19) | 8 (16)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Overall (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (7)

LIMITATIONS AND CAVEATS:
Treatment length doesn't capture metabolic benefits. Unable to evaluate maintenance of initial improvements. Limited information on length of overall exposure to antipsychotic medications. No evaluation on benefit of lifestyle.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No